CLINICAL TRIAL: NCT01404611
Title: A Multicenter, Randomized, Double-Blind Clinical Trial to Assess the Efficacy and Safety of DF289 Plus DF277 Otic Solution Compared to DF289 Otic Solution and to DF277 Otic Solution in the Treatment of Acute Otitis Media With Tympanostomy Tubes (AOMT) in Pediatric Patients
Brief Title: Efficacy and Safety of DF289 Plus DF277 Otic Solution in the Treatment of Middle Ear Infections in Pediatric Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Salvat (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DF289III/10IA04
Record Dates: First submitted 2011-07-22; First posted 2011-07-28 (Estimated); Results first posted 2015-11-23 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2015-10

CONDITIONS: Acute Otitis Media
Keywords: with tubes
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- DF289 (Active Comparator): Ear drops
  Interventions: Drug: DF289
- DF277 (Active Comparator): Ear drops
  Interventions: Drug: DF277
- DF289 plus DF277 (Experimental): Ear drops
  Interventions: Drug: DF289 plus DF277

INTERVENTIONS:
Drug: DF289 — Ear drops
  Arms: DF289
Drug: DF277 — Ear drops
  Arms: DF277
Drug: DF289 plus DF277 — Ear drops
  Arms: DF289 plus DF277

SUMMARY:
The purpose of this study is to determine if a combination of an antibiotic plus a corticosteroid is safe and effective in treating middle ear infections in children with ear tubes.

ELIGIBILITY:
Inclusion Criteria:

* 6 months to 12 years
* ear tube in the ear which will be treated
* otorrhea for 3 weeks or less
* moderate or severe otorrhea

Exclusion Criteria:

* other ear diseases

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 331 (Actual)
Dates: Start 2011-06; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratorios SALVAT S.A., Esplugues de Llobregat, Barcelona, Spain

REFERENCES:
- [Derived] Spektor Z, Pumarola F, Ismail K, Lanier B, Hussain I, Ansley J, Butehorn HF 3rd, Esterhuizen K, Byers J, Douglis F, Lansford B, Hernandez FJ. Efficacy and Safety of Ciprofloxacin Plus Fluocinolone in Otitis Media With Tympanostomy Tubes in Pediatric Patients: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2017 Apr 1;143(4):341-349. doi: 10.1001/jamaoto.2016.3537. PMID 28006041

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DF289 | DF277 | DF289 Plus DF277
Started | 112 | 108 | 111
Completed | 104 | 89 | 106
Not Completed | 8 | 19 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DF289 | DF277 | DF289 Plus DF277 | Total
Number analyzed (Participants) | 112 | 108 | 111 | 331
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 112 | 108 | 111 | 331
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.3 (2.4) | 3.2 (2.3) | 3.2 (2.5) | 3.2 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 49 | 46 | 138
  Male | 69 | 59 | 65 | 193

OUTCOME MEASURES:

1. Primary Outcome: Time to Cessation of Otorrhea
Time Frame: From baseline until the end of the study (up to 22 days)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | DF289 | DF277 | DF289 Plus DF277
Number analyzed (Participants) | 112 | 108 | 111
days | 6.83 [5.49 to 7.74] | 22 [13.93 to 22] | 4.94 [3.74 to 5.52]

ADVERSE EVENTS:
Time Frame: During all the study (22 days)
Description: There were 331 patients randomized in the study, but only 330 patients were dosed. Only dosed patients are considered for the Adverse Event Reporting.
Arm/Group | DF289 | DF277 | DF289 Plus DF277
Serious Adverse Events (participants affected / at risk) | 1/112 | 0/107 | 1/111
Other Adverse Events (participants affected / at risk) | 20/112 | 29/107 | 25/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DF289 (N=112) | DF277 (N=107) | DF289 Plus DF277 (N=111)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Non related TEAE
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Non related TEAE
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DF289 (N=112) | DF277 (N=107) | DF289 Plus DF277 (N=111)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 7 (7) — Non related TEAE
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 6 (6) | 6 (6) — Non related TEAE
Nasopharyngitis (Infections and infestations) | 1 (1) | 6 (7) | 1 (1) — Non related TEAE
Otorrhoea (Ear and labyrinth disorders) | 7 (8) | 7 (7) | 6 (6) — Only 1 event in the DF289 group and 2 events in the DF277 group were considered related TEAE. The other events were considered non related TEAE
Pyrexia (General disorders) | 8 (8) | 14 (14) | 10 (10) — Non related TEAE

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor does not object to publication by Institution of the results of the Trial based on information collected or generated by Institution, whether or not the results are favorable to the Sponsor Drug. However, to ensure against inadvertent disclosure of Confidential Information or unprotected Inventions, Institution will provide Sponsor an opportunity to review any proposed publication or other type of disclosure before it is submitted or otherwise disclosed.